CLINICAL TRIAL: NCT02623751
Title: Phase 1 Study of KHK2375 in Subjects With Advanced or Recurrent Breast Cancer
Brief Title: Study of KHK2375 in Subjects With Advanced or Recurrent Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2375-001
Record Dates: First submitted 2015-11-18; First posted 2015-12-08 (Estimated); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — exemestane; entinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- KHK2375 PO and Exemestane PO (Experimental): KHK2375 and Exemestane
  Interventions: Drug: KHK2375; Drug: Exemestane

INTERVENTIONS:
Drug: KHK2375 — KHK2375 will be orally administered once weekly. KHK2375 in combination with exemestane will be repeatedly administered in a 28-day cycle.
  Exemestane will be orally administered once daily.
Drug: Exemestane — KHK2375 will be orally administered once weekly. KHK2375 in combination with exemestane will be repeatedly administered in a 28-day cycle.
  Exemestane will be orally administered once daily.
  Other Names: Entinostat; MS-275; SDNX-275

SUMMARY:
The primary objective of the open-label, dose-escalation study is to investigate the safety of single-dose monotherapy and repeated-dose of KHK2375 combined with exemestane in female subjects with advanced or recurrent breast cancer. The secondary objective is to investigate the pharmacokinetics and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women aged ≥ 20 and < 75 years at the time of consent;
* Estrogen receptor positive and/or progesterone receptors positive;
* HER2-negative
* Nonresectable advanced or recurrent breast cancer previously treated with nonsteroidal aromatase inhibitor (AI), and planning to be treated with exemestane

Exclusion Criteria:

* Radiation therapy or immuno therapy within 14 days before the first dose of investigational product;
* Chemotherapy, biological medicines, other pharmacotherapy or major surgery within 21 days before the first dose of the investigational product;
* Prior chemotherapies of ≥ 3 regimens for advanced or recurrent breast cancer;
* Ongoing treatment with other investigational product

Ages: 20 Years to 74 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2020-10 (Actual); Study Completion 2020-10 (Actual)

PRIMARY OUTCOMES:
Number and percentage of subjects with treatment-emergent adverse events including dose-limiting toxicities and serious adverse events | Assessed up to 28 days after study discontinuation

SECONDARY OUTCOMES:
Pharmacokinetics of KHK2375 [maximum concentration (Cmax)] | Pre-dose, Cycle 0 Days 1, 2, 4, 6, Cycle 1 Days 1, 2, 4, 6, 8, 15, 22 and Cycle 2 Day 1
Pharmacokinetics of KHK2375 [Area under the curve (AUC)] | Pre-dose, Cycle 0 Days 1, 2, 4, 6, Cycle 1 Days 1, 2, 4, 6, 8, 15, 22 and Cycle 2 Day 1
Pharmacokinetics of KHK2375 [Half-life (t1/2)] | Pre-dose, Cycle 0 Days 1, 2, 4, 6, Cycle 1 Days 1, 2, 4, 6, 8, 15, 22 and Cycle 2 Day 1

CONTACTS AND LOCATIONS:
Locations (3):
- Japan (3):
  - Chikusa-ku, Aichi-ken
  - Chuo-ku, Osaka
  - Chuo-ku, Tokyo

REFERENCES:
- [Derived] Masuda N, Tamura K, Yasojima H, Shimomura A, Sawaki M, Lee MJ, Yuno A, Trepel J, Kimura R, Nishimura Y, Saji S, Iwata H. Phase 1 trial of entinostat as monotherapy and combined with exemestane in Japanese patients with hormone receptor-positive advanced breast cancer. BMC Cancer. 2021 Nov 24;21(1):1269. doi: 10.1186/s12885-021-08973-4. PMID 34819039